CLINICAL TRIAL: NCT04644549
Title: Natural History Study of Batten Disease
Status: Terminated | Type: Observational
Why Stopped: study terminated following strategic portfolio and R&D alignment
Sponsor: Emily de los Reyes (Other)
Responsible Party: Sponsor-Investigator, Emily de los Reyes, Sponsor-Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: BAT-001
Record Dates: First submitted 2020-10-27; First posted 2020-11-25 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Batten Disease; Neuronal Ceroid Lipofuscinosis CLN6; Neuronal Ceroid Lipofuscinosis CLN3
Keywords: Neuronal ceroid lipofuscinosis (NCL); CLN6; vLINCL6; CLN6 Batten Disease; Batten Disease; CLN3; CLN3 Batten Disease; variant late infantile
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Subjects with CLN6 Batten disease
- Subjects with juvenile CLN3 Batten disease

SUMMARY:
This is a multicenter, international, study to assess the natural history data from people with Batten disease by collecting both retrospective and prospective information about the motor, behavioral and functional capabilities of patients. The study initially has 2 cohorts. Cohort 1 (n ≈ 75) includes subjects with CLN6 Batten disease. Cohort 2 (n ≈ 120) includes subjects with juvenile CLN3 Batten disease. Additional cohorts for other Batten disease subtypes may be added in the future.

ELIGIBILITY:
Inclusion Criteria:

* Subject has or had a diagnosis of CLN6 or CLN3 Batten disease that has been confirmed by genotyping (documented presence of a variant on both gene alleles). Confirmation of genotyping will be performed prior to enrollment.
* Subject (or legally authorized representative) has provided written informed consent (or assent) and authorization for use and disclosure of personal health information or research related health information
* Subjects may enroll starting from birth

Exclusion Criteria:

* Subject has or had experienced another illness that is known to cause cognitive decline (eg, trauma, meningitis, hemorrhage)
* Subject received or receives an investigational gene therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects diagnosed with CLN3 or CLN6 and their parents/legal guardians are eligible to take part in this study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Assess the change over time in rating as determined using the Unified Batten Disease Rating Scale (UBDRS). | 10 years
  The UBDRS is a clinical ratings instrument used specifically to assess motor, seizure, behavioral and functional capabilities.
Assess the change over time in rating as determined using the Hamburg Scale. | 10 years
  The Hamburg scale is an established tool to capture the rate of decline or regression.
Assess the change over time in cognitive function using Mullen Scales of Early Learning (for children up to 60 months old). | 10 years
Assess the change over time in cognitive function using WPPSI-IV (for children up to 7 years 7 months old). | 10 years
Assess the change over time in cognitive function using WISC-V (for patients older than 6 years old). | 10 years
Characterize the age of onset of disease, including the timing of both the loss of capacities and the emergence of disease-related signs and symptoms | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States